CLINICAL TRIAL: NCT01217567
Title: Subcuticular Suture Versus Staples for Closure of the Skin After Caesarean Section: A Prospective Randomized Single-blinded Case-Control Study With the Case as it's Own Control.
Brief Title: Subcuticular Suture Versus Staples for Closure of the Skin After Caesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: University of Copenhagen (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Anna Aabakke, Anna Aabakke, M.D., Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cicatricestudiet; SJ-162 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Cesarean Section; Cicatrix
Keywords: cicatrix; cesarean section; sutures; surgical staples; postoperative pain; Infection
MeSH Terms: conditions — Cicatrix; Pain, Postoperative; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1st c-section, no previous lower abdominal surgery - s.l. (Experimental)
  Interventions: Procedure: Staples left, subcuticular suture right
- Woman with previous ceasarean section - staples left (Experimental)
  Interventions: Procedure: Staples left, subcuticular suture right
- 1st c-section, no previous lower abdominal surgery (Experimental)
  Interventions: Procedure: Subcuticular suture left side and staples right
- Woman with previous ceasarean section (Experimental)
  Interventions: Procedure: Subcuticular suture left side and staples right

INTERVENTIONS:
Procedure: Staples left, subcuticular suture right — Closure of the skin after cesarean section with staples on the left side of the wound and subcuticular suture on the right side.
  Arms: 1st c-section, no previous lower abdominal surgery - s.l.; Woman with previous ceasarean section - staples left
Procedure: Subcuticular suture left side and staples right — Closure of the skin after cesarean section with staples on the right side of the wound and subcuticular suture on the left side.
  Arms: 1st c-section, no previous lower abdominal surgery; Woman with previous ceasarean section

SUMMARY:
The Purpose of this study is to compare two methods for closure of the skin after caesarean section on the same patient; staples and subcuticular sutures. The study is performed on two separate groups of patients: 1. Woman having cesarean section for the first time and have not previously had abdominal surgery through a lower abdominal transverse incision. 2. Woman, who have previously had a caesarean section done. The following parameters are registered:

1. An objective evaluation of the two ends of the scar 6 months postoperatively.
2. A patient evaluation of the two ends of the scar 6 months postoperatively.
3. The difference in pain in the two ends of the scar 1 day postoperatively (blinded).
4. The difference in pain in the two ends of the scar 7 days, 3 and 6 months postoperatively.
5. The rate of infection.

ELIGIBILITY:
Inclusion Criteria:

* Woman having elective or level III caesarean section. Level III caesarean section is defined as being ordered more than 30 minutes before surgery is started.
* Woman who speak and understand Danish
* Woman who can give informed consent.

Exclusion Criteria:

* Level I or II caesarean section (ordered less than 30 min. before surgery is started).
* Diabetics (this does not include gestational diabetes).
* Infection
* Regular treatment with immunosuppressives
* Alcohol or drug abuse
* Age under 18
* Chronic pain disease eg fibromyalgia, rheumatoid arthritis
* BMI over 35
* Previous abdominal surgery through lower transverse abdominal incision (only applicable to woman having caesarean section for the first time).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Preferred side of the caesarean section scar | 6 months postoperatively
  Preferred side of the scar and thereby method for closure of the skin: Staples, subcuticular suture or no difference.

SECONDARY OUTCOMES:
The difference in pain between the two ends of the scar | 1 and 7 days postoperatively
  Difference in painscore between the two ends of the scar 1st and 7th postoperative day. Pain is registered by a score on a vas-scale from 0-10.
The difference in pain between the two ends of the scar | 3 and 6 months postoperatively
  Difference in painscore between the two ends of the scar 3 and 6 months postoperatively. Pain is registered by a score on a vas-scale from 0-10.
Pain in the two ends of the scar | 1 and 7 days postoperatively
  Pain in the two ends of the scar registered by a score on a vas-scale from 0-10 1 and 7 days postoperatively.
Pain in the two ends of the scar | 3 and 6 months postoperatively
  Pain in the two ends of the scar registered by a score on a vas-scale from 0-10 3 and 6 months postoperatively.
Infection | 7 days postoperatively
  The rate of postoperative infection and what side of the scar - right or left -that is infected.
Infection | 3 and 6 months postoperatively
  The rate of postoperative infection and what side of the scar - right or left -that is infected.
Cosmetic objective evaluation of the two ends of the scar | 6 months postoperatively
  Evaluation of the right and left side of the scar respectively by two blinded doctors using the Singer's "scar evaluation scale" . Difference in Singer's score between the two ends of the scar.
Comparison of outcome measures in woman with no previous abdominal surgery and woman with previous caesarean section. | 6 months
  Primay and Secondary outcome measures are compared in the two groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jørgen Secher, Profesoor, M.D., Study Chair — Department of Obstetrics, Hvidovre Hospital; Anna J. M. Aabakke, M.D., Principal Investigator — Department of Gynaechology and Obstetrics, Holbæk Sygehus
Locations (1):
- Department of Gynaechology and Obstetrics, Holbæk Sygehus, Holbæk, Denmark

REFERENCES:
- [Background] The CAESAR study: http://www.npeu.ox.ac.uk/caesar
- [Background] Jenkins TR. It's time to challenge surgical dogma with evidence-based data. Am J Obstet Gynecol. 2003 Aug;189(2):423-7. doi: 10.1067/s0002-9378(03)00587-8. PMID 14520211
- [Background] CORONIS Trial Collaborative Group. The CORONIS Trial. International study of caesarean section surgical techniques: a randomised fractional, factorial trial. BMC Pregnancy Childbirth. 2007 Oct 22;7:24. doi: 10.1186/1471-2393-7-24. PMID 18336721
- [Background] Altman AD, Allen VM, McNeil SA, Dempster J. Pfannenstiel incision closure: a review of current skin closure techniques. J Obstet Gynaecol Can. 2009 Jun;31(6):514-520. doi: 10.1016/S1701-2163(16)34213-X. PMID 19646316
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Gaertner I, Burkhardt T, Beinder E. Scar appearance of different skin and subcutaneous tissue closure techniques in caesarean section: a randomized study. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):29-33. doi: 10.1016/j.ejogrb.2007.07.003. Epub 2007 Sep 6. PMID 17825472
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Background] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Background] Alderdice F, McKenna D, Dornan J. Techniques and materials for skin closure in caesarean section. Cochrane Database Syst Rev. 2003;(2):CD003577. doi: 10.1002/14651858.CD003577. PMID 12804476
- [Background] Johnson A, Young D, Reilly J. Caesarean section surgical site infection surveillance. J Hosp Infect. 2006 Sep;64(1):30-5. doi: 10.1016/j.jhin.2006.03.020. Epub 2006 Jul 5. PMID 16822582
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Derived] Aabakke AJM, Krebs L, Pipper CB, Secher NJ. Subcuticular suture compared with staples for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Oct;122(4):878-884. doi: 10.1097/AOG.0b013e3182a5f0c3. PMID 24084548